CLINICAL TRIAL: NCT05473364
Title: Acetazolamide and Tubuloglomerular Feedback in Persons With Type 1 Diabetes: A Dose Finding Clinical Trial
Brief Title: Acetazolamide in Persons With Type 1 Diabetes - Dose Finding
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Assistant Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UC-MEDJP-05
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: acetazolamide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Escalating dose finding trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetazolamide - 62.5mg Dose (Experimental): 2-week treatment period with 62.5mg dose of acetazolamide taken twice daily.
  Interventions: Drug: Acetazolamide
- Acetazolamide - 125mg Dose (Experimental): 2-week treatment period with 125mg dose of acetazolamide taken twice daily.
  Interventions: Drug: Acetazolamide
- Acetazolamide - 250mg Dose (Experimental): 2-week treatment period with 250mg dose of acetazolamide taken twice daily.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Diuretic and carbonic anhydrase inhibitor medication

SUMMARY:
This is a dose finding trial where participants will receive escalating doses of acetazolamide, each for a 2-week dosing period followed by a 2-week washout period. The three doses examined will be open-label 62.5mg twice daily, 125mg twice daily, and 250mg twice daily of acetazolamide. A baseline Iohexol GFR (glomerular filtration rate) measurement will be performed prior to the first administration of each acetazolamide dose and then again following each dosing period. Including a screening visit and a follow-up visit, there will be a total of 8 study visits over approximately 16 weeks.

DETAILED DESCRIPTION:
Open-label acetazolamide will be given to persons with type 1 diabetes to determine the optimal dose to be used in a dose finding trial design. Each dose of acetazolamide will be given for a 2-week period, followed by a 2-week washout period. The three doses examined will be open-label 62.5mg twice daily, 125mg twice daily, and 250mg twice daily of acetazolamide.

To measure mGFR (measured glomerular filtration rate), an Iohexol GFR procedure will be completed at the beginning and end of each treatment period. We will follow a standard protocol for the procedure that has been used in multiple studies. Iohexol (Omnipaque 300®) will be used in order to obtain a precise measure of mGRF throughout the course of the test. Iohexol will be prepared by the UCSD (University of California, San Diego) Investigational Drug Services at the ACTRI (Altman Clinical and Translation Research Institute) by drawing up 5mL into a syringe per standard pharmacy protocol. The iohexol will be dispensed to a nurse or research coordinator who will weigh the syringe prior to infusion and again after infusion to assess exact dosage delivered.

A study nurse will insert 1 IV (intravenous) line in the hand or arm for the infusion of iohexol. They will then insert a second IV in the opposite arm for blood collection. Serial blood draws will occur throughout the procedure relative to the time of iohexol infusion. A study nurse will infuse iohexol over a 1-2 minute period, flush with 10mL of normal saline and remove the IV. Blood samples will be collected at the following time points for mGFR analysis:

* -5 minutes (prior to iohexol infusion)
* 2 hours (120 minutes post infusion)
* 4 hours (120 minutes post infusion)
* 6 hours (120 minutes post infusion)

Following completion and analysis of the dose finding trial, the optimal dose of acetazolamide will be chosen for a crossover trial based on the largest mean reduction in mGFR while avoiding a significant median reduction in sodium bicarbonate and/or potassium.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ≥ 18 years at the time of consent.
2. Females of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception during the entire study.
3. Male subjects must be willing to use clinically acceptable method of contraception during the entire study.
4. Have a clinical diagnosis of Type 1 Diabetes on a stable medication regimen for at least 3 months.
5. eGFR (estimated glomerular filtration rate) ≥ 45ml/min/1.73m2
6. Serum bicarbonate ≥ 24 meq/L
7. Negative urine toxicology screen.
8. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History of allergic reaction to acetazolamide, another carbonic anhydrase inhibitor, or any of the inactive ingredients in the acetazolamide tablets.
2. Liver disease (clinical diagnosis of cirrhosis by imaging of physician; > 14 drinks/week; AST (aspartate aminotransferase), ALT (alanine aminotransferase), or total bilirubin > 2 times the upper limit of normal).
3. Serum hemoglobin A1c > 10.0%
4. Serum hemoglobin concentration of <8 g/dL.
5. Use of > 4 anti-hypertensives, or systolic blood pressure >160mm Hg at the screening visit.
6. Use of loop, thiazide or potassium sparing diuretics.
7. A medical condition requiring active surgical or medical intervention whose urgency would preclude participation in this study at the discretion of the site investigator {active cardiac or pulmonary conditions, ongoing ischemia or cardiac symptoms, uncorrected CAD (coronary artery disease) or decompensated CHF(congestive heart failure)}.
8. Institutionalized individual (prisoners, patients with signification mental illness, or nursing home residents).
9. Active pregnancy, breastfeeding, or planning to become pregnant during the study period.
10. Current participation in another clinical trial (observational studies are exempted).
11. In the opinion of the investigators, inability to adhere to the study medical regimen or comply with recommendations.
12. Inability or unwillingness to travel to study visits.
13. Life expectancy < 1 year.
14. Hospitalization within 60 days prior to screening.
15. A plan to leave the geographical area within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in mGFR percent | 2 Weeks
  The change in mGFR percent from pre-dosing to post-treatment as measured by the iohexol procedure.
Preservation of Serum Bicarbonate | 2 Weeks
  The preservation of serum bicarbonate concentrations at ≥ 22 meq/L from pre-dosing to post treatment.
Preservation of Serum Potassium | 2 Weeks
  The preservation of serum potassium concentrations at ≥ 3.2 meq/L from pre-dosing to post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ginsberg C, Seegmiller JC, Vallon V, SeungMi Jin S, Thomas RL, Boeder SC, Pettus J, Ix JH. Acetazolamide Therapy and Kidney Function in Persons with Nonalbuminuric Diabetes Mellitus Type 1. J Am Soc Nephrol. 2025 Mar 1;36(3):463-470. doi: 10.1681/ASN.0000000515. Epub 2024 Oct 8. PMID 39466253